CLINICAL TRIAL: NCT05202483
Title: A Novel Appendicitis TriMOdal Prediction Score (ATMOS) for Acute Appendicitis in Pregnancy: a Retrospective Observational Study
Acronym: ATMOS
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: Goran Augustin (Unknown); Ognjen Barcot (Unknown); Mislav Herman (Unknown); Salvatore Giovanni Vitale (Unknown)
Responsible Party: Principal Investigator, Branko Bogdanic, MD, PhD, Clinical Hospital Centre Zagreb
Other Study IDs: 202101
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Appendicitis in Pregnancy
Keywords: appendicitis, pregnancy, score, ultrasound, neutrophil-lymphocyte ratio, CRP-platelet ratio
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute appendicitis (AA) is a disease of younger age, but it occurs in 1 out of 500-2000 pregnancies. The current treatment of choice for AA in pregnancy is surgical. Even with standard clinical examination, serum inflammatory markers, and transabdominal ultrasound, the decision on surgical treatment of acute appendicitis (AA) and the rate of negative appendectomy in pregnancy are still unsatisfactory. There are several scoring systems (Alvarado, Tzanakis) that help making decision on operating more easier, however their specificity is either high with low sensitivity, or the other way around. In addition, all scores are based on adult non-pregnant population. We are making an observational study to develop a scoring system that would include ultrasonic imaging with clinical-biochemical parameters while not compromising sensitivity and specificity.

DETAILED DESCRIPTION:
The study includes extraction of medical data for pregnant women, age 18 years or older, admitted to the University Hospital Centre Zagreb, Zagreb, Croatia, with the suspicion of AA, from January 2010 to December 2020. The aim of this study is to develop a scoring system that would include ultrasonic imaging with clinical-biochemical parameters while not compromising sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women, age 18 years or older, admitted to the University Hospital Centre Zagreb, Zagreb, Croatia, with the suspicion of acute appendicitis, from January 2010 to December 2020.

Exclusion Criteria:

* non-pregnant patients
* pregnant patients younger than 18 years
* diagnosis made with CT or MRI
* pregnant patients with the acute abdomen (intraoperative diffuse peritonitis) from acute appendicitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients (pregnant women, age 18 years or older, admitted to the University Hospital Centre Zagreb, Zagreb, Croatia, with the suspicion of acute appendicitis, from January 2010 to December 2020.) demographics, symptoms, laboratory findings, diagnostic and treatment modalities were extracted from electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Predictive factors of acute appendicitis in pregnancy | January 2010 to December 2020
  Detection of predictive factors of acute appendicitis in pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Zagreb, Zagreb, Croatia

REFERENCES:
- [Background] Golz RA, Flum DR, Sanchez SE, Liu X, Donovan C, Drake FT. Geographic Association Between Incidence of Acute Appendicitis and Socioeconomic Status. JAMA Surg. 2020 Apr 1;155(4):330-338. doi: 10.1001/jamasurg.2019.6030. PMID 32129808
- [Background] Augustin G, Majerovic M. Non-obstetrical acute abdomen during pregnancy. Eur J Obstet Gynecol Reprod Biol. 2007 Mar;131(1):4-12. doi: 10.1016/j.ejogrb.2006.07.052. Epub 2006 Sep 18. PMID 16982130
- [Background] Di Saverio S, Podda M, De Simone B, Ceresoli M, Augustin G, Gori A, Boermeester M, Sartelli M, Coccolini F, Tarasconi A, De' Angelis N, Weber DG, Tolonen M, Birindelli A, Biffl W, Moore EE, Kelly M, Soreide K, Kashuk J, Ten Broek R, Gomes CA, Sugrue M, Davies RJ, Damaskos D, Leppaniemi A, Kirkpatrick A, Peitzman AB, Fraga GP, Maier RV, Coimbra R, Chiarugi M, Sganga G, Pisanu A, De' Angelis GL, Tan E, Van Goor H, Pata F, Di Carlo I, Chiara O, Litvin A, Campanile FC, Sakakushev B, Tomadze G, Demetrashvili Z, Latifi R, Abu-Zidan F, Romeo O, Segovia-Lohse H, Baiocchi G, Costa D, Rizoli S, Balogh ZJ, Bendinelli C, Scalea T, Ivatury R, Velmahos G, Andersson R, Kluger Y, Ansaloni L, Catena F. Diagnosis and treatment of acute appendicitis: 2020 update of the WSES Jerusalem guidelines. World J Emerg Surg. 2020 Apr 15;15(1):27. doi: 10.1186/s13017-020-00306-3. PMID 32295644
- [Background] Augustin G, Boric M, Barcot O, Puljak L. Discordant outcomes of laparoscopic versus open appendectomy for suspected appendicitis during pregnancy in published meta-analyses: an overview of systematic reviews. Surg Endosc. 2020 Oct;34(10):4245-4256. doi: 10.1007/s00464-020-07674-6. Epub 2020 Jun 16. PMID 32556754
- [Background] Yang J, Wen SW, Krewski D, Corsi DJ, Walker M, Mattison D, Moog R, McNair D, Huang H, Zhuang G. Association of treatments for acute appendicitis with pregnancy outcomes in the United States from 2000 to 2016: Results from a multi-level analysis. PLoS One. 2021 Dec 13;16(12):e0260991. doi: 10.1371/journal.pone.0260991. eCollection 2021. PMID 34898628
- [Background] Ahmed S, Jha A, Ali FM, Ghareeb AE, Garg D, Jha M. Sensitivity and Specificity of the Neutrophil-lymphocyte Ratio in the Diagnosis of Acute Appendicitis. Ann Clin Lab Sci. 2019 Sep;49(5):632-638. PMID 31611206
- [Background] Sigdel GS, Lakhey PJ, Mishra PR. Tzanakis score vs. Alvarado score in acute appendicitis. JNMA J Nepal Med Assoc. 2010 Apr-Jun;49(178):96-9. PMID 21485591
- [Derived] Augustin G, Mikus M, Bogdanic B, Barcot O, Herman M, Goldstajn MS, Tropea A, Vitale SG. A novel Appendicitis TriMOdal prediction Score (ATMOS) for acute appendicitis in pregnancy: a retrospective observational study. Updates Surg. 2022 Dec;74(6):1933-1941. doi: 10.1007/s13304-022-01368-5. Epub 2022 Sep 1. PMID 36048362